CLINICAL TRIAL: NCT04933175
Title: Fluzopalil in Combination With Anlotinib for Extensive Small-cell Lung Cancer Following Failure of First-line Platinum-containing Chemotherapy: a Multicenter, Single-arm Prospective Phase II Clinical Study (STAMP Study)
Brief Title: Fluzopalil in Combination With Anlotinib for Extensive Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liu Zhenhua (Other)
Responsible Party: Sponsor-Investigator, Liu Zhenhua, Director, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LZhenhua
Record Dates: First submitted 2021-06-07; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: Fluzopali combined with anlotinib for extensive stage small cell lung cancer after failure of first-line platinum-containing chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fluzopali combined with anlotinib (Experimental): Patients 18 years of age or older, 75 years of age or younger with histologically proven small cell carcinoma of the lung were assessed by radiography as having an extensive stage (according to the American Veteran Lung Cancer Association). Patients received first-line two-drug chemotherapy with standard cisplatin, carboplatin, or lobaplatin, combined with or without immunotherapy, and developed radiologically evaluated disease progression during treatment or within 6 months of completion of treatment.
  Interventions: Drug: Fluzoparil; Drug: Anlotinib

INTERVENTIONS:
Drug: Fluzoparil — Fluzoparil: 150 mg, P.O, BID, d1-14, Q3W; Treatment until disease progression or intolerable side effects occur.
Drug: Anlotinib — Anlotinib: 8mg, P.O, qd, d1-14, Q3W; Treatment until disease progression or intolerable side effects occur.

SUMMARY:
This is a the researchers launched a multicenter, prospective, single arm phase II clinical study, the group always had at least two cycle line standard platinum-based treatment and curative effect for SD, at least 6 months during or after the treatment of disease progression broad stage small cell lung cancer patients, evaluating the efficacy and safety of fluzopalil combination With anlotinib. Fifty patients are expected to be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

-

To be included in the study, subjects must meet all of the following inclusion criteria:

1. Volunteered to participate in the study, signed the informed consent, had good compliance, and cooperated with follow-up;
2. Age ≥ 18 years old, ≤ 75 years old, gender is not limited;
3. Histological diagnosis of small cell lung cancer, radiographic classification according to the American Legion Lung Cancer Association is extensive stage;
4. There is at least 1 evaluable lesion according to RECIST1.1, has not received previous local treatment such as irradiation, has not received tissue biopsy during the screening phase, and can be accurately measured at baseline, maximum diameter ≥ 10 mm at baseline (short diameter ≥ 15 mm if lymph node is present). The measurement method chosen is suitable for accurate repeated measurements and can be computed tomography (CT) or magnetic resonance imaging (MRI). If there is only one measurable lesion and no prior local treatment such as irradiation, it can be accepted as the target lesion and the baseline evaluation of the tumor lesion should be performed at least 14 days after the diagnostic biopsy.
5. Patients who have received at least 2 cycles of standard platinum-containing chemotherapy (cisplatin, carboplatin or Lobaplatin) with a efficacy of at least SD and who have developed disease progression according to RECIST1.1 as assessed by imaging during treatment or within 6 months after the end of the last treatment;
6. The Eastern Cooperative Tumor Group (ECOG) physical status score was 0-2, with a minimum expected survival of 12 weeks;
7. Peripheral blood and liver and renal function within the following allowable range (detected within 7 days before the start of treatment) :

   * leukocytes (WBC) ≥3.0×109/L or neutrophils (ANC) ≥1.5×109/L;
   * hemoglobin (HGB) ≥80 g/L;
   * platelet (PLT) ≥80×109/L;
   * liver transaminase (AST, ALT) < 2.5 times of the upper limit of the normal range;
   * Total bilirubin (TBIL) < 2 times the upper limit of the normal range;
   * creatinine (CREAT) < 1.5 times the upper limit of the normal range;
8. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%);
9. Women of childbearing age should take appropriate contraceptive measures and should not breastfeed for 3 months from screening to the cessation of study treatment. Negative pregnancy test (urine or serum) within 7 days prior to the start of administration, or no risk of pregnancy if one of the following criteria is met:

A. Postmenopausal is defined as being older than 50 years of age and amenorrhea for at least 12 months after the cessation of all exogenous hormone replacement therapy; B. Women younger than 50 years of age may be considered postmenopausal if they have had amenorrhea for 12 months or more after discontinuation of all exogenous hormone therapy and their luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the laboratory postmenopausal reference range; C. Has undergone irreversible sterilization, including hysterectomy, bilateral oophorectomy or bilateral salpingectomy, except for bilateral tubal ligation; 10.Men should use barrier contraception (i.e., condoms) for 3 months from screening to discontinuation of study treatment.

Exclusion Criteria:

-

Subjects will not be enrolled in this study if they meet any of the following criteria:

1. Previous primary drug resistance to standard platinum two-drug chemotherapy;
2. Have received any of the following treatments:

   A. Previous use of any PARP inhibitors or antiangiogenic agents, including anlotinib, bevacizumab, sorafenib; B. Patients who had undergone major surgery within 4 weeks prior to the first dosing of the study drug; C. Have received more than 30% bone marrow irradiation or large area radiotherapy within 4 weeks prior to first dosing of the study drug;
3. Patients complicated with other malignant tumors, except basal cell carcinoma of the skin and carcinoma in situ;
4. Imaging (CT or MRI) showed obvious pulmonary cavitary tumor;
5. Participating in other clinical studies or participating in other clinical studies within 4 weeks prior to study commencement;
6. Known to be allergic to the study drug ingredients;
7. Within 4 weeks before the first dose of test drug treatment has received chemotherapy, radiation therapy, or other test with anticancer therapy (double phosphate except drugs) : always had received a local radiotherapy, if can meet the following conditions into groups: radiation from the end of the treatment to more than 4 weeks (brain radiotherapy for more than 2 weeks). In addition, the target lesions selected in this study were not in the radiotherapy area. Or if the target lesion is within the radiotherapy area but has been confirmed to have progressed;
8. Patients with antitumor treatment-related adverse reactions (except alopecia) that did not recover to NCI-CTCAE≤ grade 1 after previous systemic antitumor therapy;
9. Abnormal coagulation function (INR >1.5 or prothrombin time (PT) > ULN+4 s or APTT >1.5 ULN), bleeding tendency or receiving thrombolytic or anticoagulant therapy; Note: Low dose heparin (60 000 ~ 12 000 U per day for adults) or low dose aspirin (100 mg or less per day) are allowed for prophylactic purposes on the premise that INR is ≤1.5.
10. Clinically significant hemoptysis (more than half tablespoon of hemoptysis per day) occurred within 3 months before enrollment; Or 4 weeks before the group has significant clinical significance of bleeding or bleeding tendency, such as gastrointestinal bleeding, bleeding ulcers (including gastrointestinal perforation and/or fistula, but already after surgical removal of the gastrointestinal tract perforation or fistula, can be allowed into the group), baseline period + + and above of defecate occult blood, healing wounds, ulcers or fracture, etc.;
11. Renal insufficiency: Routine urine indicated that urinary protein was ≥ ++, or confirmed that the 24-hour urinary protein amount was > 1.0g;
12. Patients with unsatisfactory blood pressure control after medication (systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg);
13. Suffers from serious cardiovascular diseases: Myocardial ischemia or myocardial infarction above Ⅱ, poorly controlled arrhythmia; According to NYHA standard, Ⅲ ~ L cardiac dysfunction, or heart color ultrasound examination indicated left ventricular ejection fraction (LVEF) < 50%;
14. Peripheral neuropathy ≥CTCAE 2 is present, except due to trauma;
15. Uncontrolled medium to large serosal effusions (including pleural effusion, ascites, and pericarpericidal effusion) after pumping treatment, aggravated chronic obstructive pulmonary disease, active pulmonary infection and/or acute bacterial or fungal respiratory disease requiring intravenous antibiotic treatment;
16. Factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction;
17. Artery/venous thrombosis events, such as cerebrovascular accidents (including cerebral hemorrhage and cerebral infarction), deep venous thrombosis and pulmonary embolism, occurred within 6 months before the grouping;
18. A known history of psychotropic substance abuse, alcohol abuse or drug abuse;
19. Uncontrolled active hepatitis after treatment (hepatitis B: HBsAg positive and HBV DNA≥1 x 104 copies /ml; Hepatitis C: HCV RNA positive and abnormal liver function); Co-infection with hepatitis B and hepatitis C;
20. Women who are lactating or who have positive blood or urine pregnancy test results within 3 days before the first dosing of study therapy;
21. Patients who, as judged by the Investigator, may have poor compliance with the study procedures and requirements;
22. The investigator identified patients with any condition that jeopardized patient safety or interfered with study evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Objective Overall Response Rate (ORR) | From randomization to 24 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to 12 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
  The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.
Overall Survival (OS) | From enrollment to 24 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
  The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Disease control rate(DCR) | From enrollment to 12 month
  DCR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR or SD. DCR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR or SD to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The DCR will be reported by percentage with each arms and appropriate confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Zhuang, Dr., Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Liu Zhenhua. ZhuangWu, Fuzhou, Fujain, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li D, Huang Z, Zhong J, Lin L, Zhang G, Zhuang W, Liu Z. Efficacy and safety of fluzoparib combined with anlotinib in extensive stage small cell lung cancer after first-line platinum-based chemotherapy: a multi-center, single-arm prospective phase II clinical study (STAMP study). BMC Cancer. 2023 Aug 14;23(1):753. doi: 10.1186/s12885-023-11230-5. PMID 37580661